CLINICAL TRIAL: NCT04713319
Title: Acute Health Effects of a Bout of Exercise in Physically Active Persons and Comparison to a Repetition With Natural Signalling Agent
Brief Title: Novel Energy Metabolic Signaling Molecule With Therapeutic Potential
Acronym: RH013001
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Petteri Hirvonen (Industry)
Collaborators: University of Jyvaskyla (Other)
Responsible Party: Sponsor-Investigator, Petteri Hirvonen, Chief Scientific Officer, Replicon Health Oy
Organization: Replicon Health Oy (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019_410211_2020
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: Altogether a 25 day study with first four days non-blinded with water. There after 0-control blood samples. After the 0-control blinded treatments for 21 days (3 weeks). Study group apparently healthy 50-60 year old males and females (N=27).
Who Masked: Participant, Care Provider
Masking Description: Participants and care providers were fully blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Ten participants were randomly selected to the placebo group.
  Calcium chloride (E509) dissolved into water. Extremely small equimolar calcium dose with the test item.
  Interventions: Other: Placebo
- RH013001 (DGA) (Active Comparator): D-glyceric acid (DGA) calcium salt dehydrate (RH013001) dissolved into 1.8 dl of water. Effective dose of DGA was 3.33 mg / kg body weigh for the first 4 days. Thereafter the dose was reduced to half for the 14 days follow up period. Frequency: 2 times a day.
  Interventions: Drug: Panavital

INTERVENTIONS:
Drug: Panavital — In the morning and evening a dose of Placebo or D-glyceric acid (DGA) calcium salt dehydrate (Panavital) dissolved into 1.8 dl of water.
  Other Names: D-glyceric acid calcium salt dehydrate
  Arms: RH013001 (DGA)
Other: Placebo — In the morning and evening a dose of Placebo or D-glyceric acid (DGA) calcium salt dehydrate (Panavital) dissolved into 1.8 dl of water.
  Arms: Placebo

SUMMARY:
Altogether a 25-day study. First 4 days non-blinded with water before 0-control blood samples (Day0). Thereafter blinded for 21 days (3 weeks). Study group was apparently healthy 50-60 -year-old males and females (N=27).

DETAILED DESCRIPTION:
Blinded 21-day period was divided into two sub-periods (7 days and 14 days) and it included 3 measurement days. All measurements were on the same day of each week to facilitate maximal comparability (Day0, Day7 and Day21). Additionally on Day0 and Day7 there were acute measurements 45 minutes after morning "non-acute" resting and fasting blood samples. (In a "non-acute" measurement last dose of Panavital or placebo was taken 12 hours before the "non-acute" blood sample collected next morning .)

First week started with Day0 baseline measurements and immediately thereafter a strenuous VO2max test with 2 recovery days thereafter. After full recovery a 4-day blinded Panavital regimen. Last "non-acute" dose on Day6 was taken 12 hours before Day7 morning blood sample. At Day7 an acute 45 min placebo comparison was conducted.

Thereafter a 14-day follow-up period with halved Panavital dose or Placebo. Altogether 5 arterial blood samples were withdrawn. Three fasting and resting "non-acute" samples were taken in the morning before any treatments at Day0, Day7 and Day21. Two acute samples were collected after the VO2max (Day1) and after acute Panavital or placebo doses (Day7).

Additionally 5 fingertip blood samples for glucose (and lactate) were taken at the same time as arterial samples (Day0 and Day7) and one fingertip sample was taken immediately at the end of VO2max.

ELIGIBILITY:
Inclusion Criteria:

* healthy 50-60 year-old females and males

Exclusion Criteria:

* history of cardiovascular diseases, overweight (BMI >32)

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Acute change in blood IL-6, insulin, and glucose after RH013001 or Placebo dose at Day7 | 45 minutes control blood sample
  Immediately after morning (non-acute) blood sample therapeutic dose of RH013001 or placebo. Comparison of average response between RH013001 and placebo. Additional comparison to VO2max response (see pre-specified outcome below).
Change in blood metrices from Day1 (0-control / baseline) to Day7 | 7 days
  Last dose 12 hours earlier = "non-acute". Paired comparison to Day1, measurements included energy metabolic and anti-inflammatory markers (first 3 days for recovery from VO2max), N in blinded placebo group was 0 for the first 7 days

SECONDARY OUTCOMES:
Global RNA-sequencing | 21 days
  From 3 "non-acute" blood samples (Day1, Day7 and Day21) white blood cells collected into Paxgene tubes.
Change in "non-acute" blood sample metrices from Day1 (baseline) to Day21 | 21 days
  Intra-group paired comparison to Day1 (paired t-test of the group averages), unpaired comparison of changes in group averages between placebo and RH013001 treatment.

OTHER OUTCOMES:
Participants' Aerobic Capacity at Day1. | 10-20 + 30 minutes
  Result of the indirect maximal oxygen intake VO2max test with cycling ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Kyröläinen, PhD, Study Director — University of Jyvaskyla; Petteri Hirvonen, M.Sc., MBA, Principal Investigator — University of Jyväskylä, Replicon Health Oy
Locations (1):
- Faculty of Sports and Health Sciences, University of Jyväskylä, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: No
After deindentification of the individual data, we may share all the data that is reported in published articles. TIME FRAME: from 9 months to 36 months of the publication date. (Main data will be presented in the supplements of the articles.) Original Study Protocol and Study Plan for the Ethical Committee may also be shared. TO WHOM: researches who have been accepted by independent review committee for this purpose.